CLINICAL TRIAL: NCT01421303
Title: Work Productivity In A Cohort Of Employed Ankylosing Spondylitis Patients Treated With Etanercept
Brief Title: Work Productivity in Active Ankylosing Spondylitis (AS) Patients Treated With Enbrel.
Acronym: AS@WORK
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0881A3-4675; B1801053 (Other: Alias Study Number)
Record Dates: First submitted 2011-08-19; First posted 2011-08-22 (Estimated); Results first posted 2014-12-12 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AS patients who are working and treated with Enbrel
  Interventions: Drug: Enbrel

INTERVENTIONS:
Drug: Enbrel — Enbrel

SUMMARY:
Patients with Ankylosing spondylitis more frequently discontinue work. This study measures the impact of Enbrel on work participation.

DETAILED DESCRIPTION:
Purely descriptive

ELIGIBILITY:
Inclusion Criteria:

* Active AS patients (as judged by the treating MD) who are currently employed.
* Patients who are scheduled by their rheumatologist to initiate treatment with Etanercept.

Exclusion Criteria:

* Patients who initiated a procedure for eligibility of work disability/pension.
* Patients with previous use of TNF-alpha inhibitors either in commercial use, or in a study for the treatment of AS or a related spondylarthropathy condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AS patients visiting the rheumatologist for which the decision has been taken to prescribe Enbrel
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2009-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Universitair Ziekenhuis Gent, Ghent, Gent, Belgium

REFERENCES:
- [Derived] Boonen A, Boone C, Albert A, Mielants H. Contextual factors influence work outcomes in employed patients with ankylosing spondylitis starting etanercept: 2-year results from AS@Work. Rheumatology (Oxford). 2018 May 1;57(5):791-797. doi: 10.1093/rheumatology/kex476. PMID 29373701
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A3-4675&StudyName=Work%20Productivity%20in%20Active%20Ankylosing%20Spondylitis%20%28AS%29%20Patients%20Treated%20with%20Enbrel.%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept: Participants diagnosed with active Ankylosing Spondylitis (AS) and starting an anti-Tumor Necrosis Factor (anti-TNF) treatment with etanercept (Enbrel) 25 milligram (mg) twice weekly or 50 mg once weekly were observed prospectively for up to 2 years.
Period: Overall Study
Arm/Group | Etanercept
Started | 80
Completed | 58
Not Completed | 22
Not completed — Lost to Follow-up | 13
Not completed — Non compliance with study procedure | 1
Not completed — Other | 7
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis set (BAS) consisted of all participants enrolled in the study, who were seen at baseline and started the treatment with etanercept (Enbrel).
Arm/Group | Etanercept
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 40

OUTCOME MEASURES:

1. Primary Outcome: Work Productivity and Activity Impairment Questionnaire - Ankylosing Spondylitis (WPAI-AS) Scale Scores at Baseline
Description: WPAI-AS is 6-question participant rated questionnaire to determine the amount of absenteeism, presenteeism, work productivity loss and daily activity impairment attributable to ankylosing spondylitis for a period of 7 days prior to each visit. It yields 4 sub-scores: work time missed (absenteeism), impairment while working (presenteeism or reduced on-the-job effectiveness), overall work impairment (work productivity loss or absenteeism plus presenteeism) and activity impairment (daily activity impairment). These sub-scores are transformed to impairment percentages (range from 0 to 100), with higher numbers indicating greater impairment and less productivity.
Time Frame: Baseline
Population: Baseline analysis set (BAS) consisted of all participants enrolled in the study, who were seen at baseline and started the treatment with etanercept (Enbrel). Here 'n' signifies those participants who were evaluable for the given sub-scale items at baseline.
Measure: Mean (Standard Deviation); unit: Percentage of impairment
Arm/Group | Etanercept
Number analyzed (Participants) | 80
Percentage of impairment
  Work Time Missed (n=67) | 30.18 (40.64)
  Impairment While Working (n=55) | 49.09 (22.87)
  Overall work impairment (n=49) | 53.06 (25.67)
  Activity impairment (n=79) | 63.29 (21.47)

2. Primary Outcome: Work Productivity and Activity Impairment Questionnaire - Ankylosing Spondylitis (WPAI-AS) Scale Scores at Month 6
Description: as for outcome 1
Time Frame: Month 6
Population: Follow-up analysis set (FAS) consisted of all participants enrolled in the study, who were seen at baseline, started the treatment with etanercept and had at least 1 visit during follow-up. Here 'n' signifies those participants who were evaluable for the given sub-scale items at Month 6.
Measure: Mean (Standard Deviation); unit: Percentage of impairment
Arm/Group | Etanercept
Number analyzed (Participants) | 75
Percentage of impairment
  Work Time Missed (n=61) | 6.23 (22.55)
  Impairment While Working (n=59) | 27.97 (22.42)
  Overall work impairment (n=56) | 28.07 (23.45)
  Activity impairment (n=72) | 31.81 (24.57)

3. Primary Outcome: Work Productivity and Activity Impairment Questionnaire - Ankylosing Spondylitis (WPAI-AS) Scale Scores at Month 12
Description: as for outcome 1
Time Frame: Month 12
Population: FAS consisted of all participants enrolled in the study, who were seen at baseline, started the treatment with etanercept and had at least 1 visit during follow-up. Here 'n' signifies those participants who were evaluable for the given sub-scale items at Month 12.
Measure: Mean (Standard Deviation); unit: Percentage of impairment
Arm/Group | Etanercept
Number analyzed (Participants) | 75
Percentage of impairment
  Work Time Missed (n=55) | 5.52 (22.91)
  Impairment While Working (n=56) | 25.18 (22.40)
  Overall work impairment (n=51) | 23.97 (21.75)
  Activity impairment (n=67) | 29.55 (26.02)

4. Primary Outcome: Work Productivity and Activity Impairment Questionnaire - Ankylosing Spondylitis (WPAI-AS) Scale Scores at Month 18
Description: as for outcome 1
Time Frame: Month 18
Population: FAS consisted of all participants enrolled in the study, who were seen at baseline, started the treatment with etanercept and had at least 1 visit during follow-up. Here 'n' signifies those participants who were evaluable for the given sub-scale items at Month 18.
Measure: Mean (Standard Deviation); unit: Percentage of impairment
Arm/Group | Etanercept
Number analyzed (Participants) | 75
Percentage of impairment
  Work Time Missed (n=46) | 1.06 (7.17)
  Impairment While Working (n=45) | 24.89 (20.96)
  Overall work impairment (n=44) | 24.65 (21.69)
  Activity impairment (n=55) | 30.18 (24.30)

5. Primary Outcome: Work Productivity and Activity Impairment Questionnaire - Ankylosing Spondylitis (WPAI-AS) Scale Scores at Month 24
Description: as for outcome 1
Time Frame: Month 24
Population: FAS consisted of all participants enrolled in the study, who were seen at baseline, started the treatment with etanercept and had at least 1 visit during follow-up. Here 'n' signifies those participants who were evaluable for the given sub-scale items at Month 24.
Measure: Mean (Standard Deviation); unit: Percentage of impairment
Arm/Group | Etanercept
Number analyzed (Participants) | 75
Percentage of impairment
  Work Time Missed (n=41) | 6.31 (22.36)
  Impairment While Working (n=41) | 24.88 (20.39)
  Overall work impairment (n=38) | 25.88 (21.86)
  Activity impairment (n=56) | 30.18 (23.55)

6. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Questionnaire - Ankylosing Spondylitis (WPAI-AS) Scale Scores at Month 6 and 24
Description: WPAI: AS is 6-question participant rated questionnaire to determine the amount of absenteeism, presenteeism, work productivity loss and daily activity impairment attributable to ankylosing spondylitis (AS) for a period of 7 days prior to each visit. It yields 4 sub-scores: work time missed (absenteeism), impairment while working (presenteeism), overall work impairment (work productivity) and activity impairment (daily activity impairment). These sub-scores are transformed to impairment percentages (range from 0 to 100), with higher numbers indicating greater impairment and less productivity.
Time Frame: Baseline, Month 6, Month 24
Population: FAS consisted of all participants enrolled in the study, who were seen at baseline, started the treatment with etanercept and had at least 1 visit during follow-up. Here 'n' signifies those participants who were evaluable at the specified time points for the given sub-scale items.
Measure: Mean (Standard Deviation); unit: Percentage of impairment
Arm/Group | Etanercept
Number analyzed (Participants) | 75
Percentage of impairment
  Month 6: Work Time Missed (n=55) | -22.61 (40.36)
  Month 6: Impairment While Working (n=44) | -22.05 (24.55)
  Month 6: Overall work impairment (n=38) | -24.68 (27.70)
  Month 6: Activity impairment (n=72) | -31.53 (26.41)
  Month 24: Work Time Missed (n=36) | -27.11 (45.41)
  Month 24: Impairment While Working (n=27) | -29.63 (19.71)
  Month 24: Overall work impairment (n=23) | -33.44 (22.83)
  Month 24: Activity impairment (n=56) | -33.75 (25.05)

7. Secondary Outcome: Correlation Between Work Productivity and Activity Impairment Questionnaire - Ankylosing Spondylitis (WPAI-AS) Scale Scores and Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Total Score at Baseline
Description: WPAI-AS: 6-question participant rated questionnaire to determine amount of absenteeism, presenteeism, work productivity loss, daily activity impairment attributable to AS for a period of 7 days prior to each visit. It yields 4 sub-scores: work time missed (absenteeism), impairment while working (presenteeism), overall work impairment (work productivity), activity impairment (daily activity impairment). These sub-scores are transformed to impairment percentages (range from 0 to 100), with higher numbers indicating greater impairment and less productivity. BASDAI: validated self-assessment tool to determine disease activity in participants with AS. Utilizing a scale of 0-10 (0=none and 10=very severe), participants answered 6 questions measuring discomfort, pain, fatigue. The BASDAI total score averages the individual assessments and ranges from 0-10 (0=none, 10=very severe). Correlation coefficient between WPAI-AS and BASDAI score at baseline was reported.
Time Frame: Baseline
Population: BAS consisted of all participants enrolled in the study, who were seen at baseline and started the treatment with etanercept (Enbrel). Here 'n' signifies those participants who were evaluable for the given scale item at baseline.
Measure: Number; unit: Correlation coefficient
Arm/Group | Etanercept
Number analyzed (Participants) | 80
Correlation coefficient
  Work Time Missed and BASDAI (n=66) | 0.21
  Impairment While Working and BASDAI (n=55) | 0.60
  Overall work impairment and BASDAI (n=49) | 0.62
  Activity impairment and BASDAI (n=78) | 0.62

8. Secondary Outcome: Correlation Between Work Productivity and Activity Impairment Questionnaire - Ankylosing Spondylitis (WPAI-AS) Scale Scores and Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Total Score at Month 6 and Month 24
Description: WPAI-AS: 6-question participant rated questionnaire to determine amount of absenteeism, presenteeism, work productivity loss, daily activity impairment attributable to AS for a period of 7 days prior to each visit. It yields 4 sub-scores: work time missed (absenteeism), impairment while working (presenteeism), overall work impairment (work productivity), activity impairment (daily activity impairment). These sub-scores are transformed to impairment percentages (range from 0 to 100), with higher numbers indicating greater impairment and less productivity. BASDAI: validated self-assessment tool to determine disease activity in participants with AS. Utilizing a scale of 0-10 (0=none and 10=very severe), participants answered 6 questions measuring discomfort, pain, fatigue. The BASDAI total score averages the individual assessments and ranges from 0-10 (0=none, 10=very severe). Correlation coefficient between change from baseline in WPAI-AS and BASDAI score at Month 6 and 24 was reported.
Time Frame: Month 6, Month 24
Population: as for outcome 6
Measure: Number; unit: Correlation coefficient
Arm/Group | Etanercept
Number analyzed (Participants) | 75
Correlation coefficient
  Month 6: Work Time Missed and BASDAI (n=55) | 0.23
  Month 6: Impairment While Working and BASDAI(n=44) | 0.62
  Month 6: Overall work impairment and BASDAI(n= 38) | 0.56
  Month 6: Activity impairment and BASDAI (n=72) | 0.55
  Month 24: Work Time Missed and BASDAI (n=36) | 0.41
  Month 24:Impairment While Working and BASDAI(n=27) | 0.42
  Month 24:Overall work impairment and BASDAI(n= 23) | 0.40
  Month 24: Activity impairment and BASDAI (n=56) | 0.63

9. Secondary Outcome: Correlation Between Work Productivity and Activity Impairment Questionnaire - Ankylosing Spondylitis (WPAI-AS) Scale Scores and Bath Ankylosing Spondylitis Functional Index (BASFI) Total Score at Baseline
Description: WPAI-AS:6-question participant rated questionnaire to determine amount of absenteeism, presenteeism, work productivity loss, daily activity impairment due to AS for a period of 7 days prior to each visit. It yields 4 sub-scores: work time missed(absenteeism), impairment while working(presenteeism), overall work impairment(work productivity), activity impairment(daily activity impairment). These sub-scores are transformed to impairment percentages(range 0 to 100), with higher numbers indicating greater impairment, less productivity. BASFI:validated self-assessment tool to determine degree of functional limitation in AS. Utilizing a scale of 0-10(0=easy, 10=impossible),participants answered 10 questions assessing ability in completing normal daily activities/physically demanding activities. BASFI total score=mean score of 10 questions (range: 0 to 10, higher score=more severity). Correlation coefficient between WPAI-AS and BASFI score at baseline was reported.
Time Frame: Baseline
Population: as for outcome 7
Measure: Number; unit: Correlation coefficient
Arm/Group | Etanercept
Number analyzed (Participants) | 80
Correlation coefficient
  Work Time Missed and BASFI (n=67) | 0.29
  Impairment While Working and BASFI (n=55) | 0.59
  Overall work impairment and BASFI (n= 49) | 0.58
  Activity impairment and BASFI (n=79) | 0.54

10. Secondary Outcome: Correlation Between Work Productivity and Activity Impairment Questionnaire - Ankylosing Spondylitis (WPAI-AS) Scale Scores and Bath Ankylosing Spondylitis Functional Index (BASFI) Total Score at Month 6 and 24
Description: WPAI-AS:6-question participant rated questionnaire to determine amount of absenteeism, presenteeism, work productivity loss, daily activity impairment due to AS for a period of 7 days prior to each visit. It yields 4 sub-scores: work time missed(absenteeism), impairment while working(presenteeism), overall work impairment(work productivity), activity impairment(daily activity impairment). These sub-scores are transformed to impairment percentages(range 0 to 100), with higher numbers indicating greater impairment, less productivity. BASFI:validated self-assessment tool to determine degree of functional limitation in AS. Utilizing a scale of 0-10(0=easy, 10=impossible),participants answered 10 questions assessing ability in completing normal daily activities/physically demanding activities. BASFI total score=mean score of 10 questions (range: 0 to 10, higher score=more severity). Correlation coefficient between change from baseline in WPAI-AS and BASFI score at Month 6, 24 was reported.
Time Frame: Month 6, Month 24
Population: FAS consisted of all participants enrolled in the study, who were seen at visit 1 (baseline), started the treatment with etanercept and had at least one visit during follow-up. Here 'n' signifies those participants who were evaluable at specified time points for the given sub-scale items.
Measure: Number; unit: Correlation coefficient
Arm/Group | Etanercept
Number analyzed (Participants) | 75
Correlation coefficient
  Month 6: Work Time Missed and BASFI (n=55) | 0.36
  Month 6:Impairment While Working and BASFI(n=44) | 0.56
  Month 6: Overall work impairment and BASFI(n=38) | 0.62
  Month 6: Activity impairment and BASFI (n=71) | 0.62
  Month 24: Work Time Missed and BASFI (n=36) | 0.37
  Month 24:Impairment While Working and BASFI(n=27) | 0.47
  Month 24: Overall work impairment and BASFI(n=23) | 0.43
  Month 24: Activity impairment and BASFI (n=56) | 0.57

11. Secondary Outcome: Correlation Between Work Productivity and Activity Impairment Questionnaire - Ankylosing Spondylitis (WPAI-AS) Scale Scores and Bath Ankylosing Spondylitis Metrology Index (BASMI) Total Score at Baseline
Description: WPAI-AS:6-question participant rated questionnaire to determine amount of absenteeism, presenteeism, work productivity loss, daily activity impairment due to AS for a period of 7 days prior to each visit. It yields 4 sub-scores: work time missed(absenteeism), impairment while working(presenteeism), overall work impairment(work productivity), activity impairment(daily activity impairment). These sub-scores are transformed to impairment percentages(range 0 to 100), with higher numbers indicating greater impairment, less productivity. BASMI is an objective measure of spinal mobility. The BASMI score is composed of 5 measures: cervical rotation, intermalleolar distance, modified Schober's test, lateral flexion and tragus to wall distance. Final score ranges from 0 to 10: the higher the BASMI score, the more severe the participant's limitation of movement due to their AS. Correlation coefficient between WPAI-AS and BASMI score at baseline was reported.
Time Frame: Baseline
Population: as for outcome 7
Measure: Number; unit: Correlation coefficient
Arm/Group | Etanercept
Number analyzed (Participants) | 80
Correlation coefficient
  Work Time Missed and BASMI (n=65) | 0.06
  Impairment While Working and BASMI (n=53) | 0.30
  Overall work impairment and BASMI (n= 47) | 0.23
  Activity impairment and BASMI (n=77) | 0.08

12. Secondary Outcome: Correlation Between Work Productivity and Activity Impairment Questionnaire - Ankylosing Spondylitis (WPAI-AS) Scale Scores and Bath Ankylosing Spondylitis Metrology Index (BASMI) Total Score at Month 6 and 24
Description: WPAI-AS:6-question participant rated questionnaire to determine amount of absenteeism, presenteeism, work productivity loss, daily activity impairment due to AS for a period of 7 days prior to each visit. It yields 4 sub-scores: work time missed(absenteeism), impairment while working(presenteeism), overall work impairment(work productivity), activity impairment(daily activity impairment). These sub-scores are transformed to impairment percentages(range 0 to 100), with higher numbers indicating greater impairment, less productivity. BASMI is an objective measure of spinal mobility. The BASMI score is composed of 5 measures: cervical rotation, intermalleolar distance, modified Schober's test, lateral flexion and tragus to wall distance. Final score ranges from 0 to 10: the higher the BASMI score, the more severe the participant's limitation of movement due to their AS. Correlation coefficient between change from baseline in WPAI-AS and BASMI score at Month 6, 24 was reported.
Time Frame: Month 6, Month 24
Population: as for outcome 6
Measure: Number; unit: Correlation coefficient
Arm/Group | Etanercept
Number analyzed (Participants) | 75
Correlation coefficient
  Month 6: Work Time Missed and BASMI (n=50) | 0.17
  Month 6: Impairment While Working and BASMI(n=41) | 0.26
  Month 6: Overall work impairment and BASMI (n=35) | 0.12
  Month 6: Activity impairment and BASMI (n=66) | 0.31
  Month 24: Work Time Missed and BASMI (n=33) | -0.088
  Month 24: Impairment While Working and BASMI(n=24) | 0.34
  Month 24: Overall work impairment and BASMI(n=20) | 0.39
  Month 24: Activity impairment and BASMI (n=53) | -0.070

13. Secondary Outcome: Correlation Between Work Productivity and Activity Impairment Questionnaire - Ankylosing Spondylitis (WPAI-AS) Scale Scores and Bath Ankylosing Spondylitis Global Score (BAS-G) at Baseline
Description: WPAI-AS:6-question participant rated questionnaire to determine amount of absenteeism, presenteeism, work productivity loss, daily activity impairment due to AS for a period of 7 days prior to each visit. It yields 4 sub-scores: work time missed(absenteeism), impairment while working(presenteeism), overall work impairment(work productivity), activity impairment(daily activity impairment). These sub-scores are transformed to impairment percentages(range 0 to 100), with higher numbers indicating greater impairment, less productivity. BAS-G is used to indicate the effect of disease on participant's well-being. This scale is composed of 2 items ranging from 0 = very good to 10 =very bad. Total score ranges from 0 to 10: the higher the BAS-G score, the worse the participant's health status. Correlation coefficient between WPAI-AS and BAS-G score at baseline was reported.
Time Frame: Baseline
Population: as for outcome 7
Measure: Number; unit: Correlation coefficient
Arm/Group | Etanercept
Number analyzed (Participants) | 80
Correlation coefficient
  Work Time Missed and BAS-G (n=67) | 0.21
  Impairment While Working and BAS-G (n=55) | 0.48
  Overall work impairment and BAS-G (n=49) | 0.48
  Activity impairment and BAS-G (n=79) | 0.61

14. Secondary Outcome: Correlation Between Work Productivity and Activity Impairment Questionnaire - Ankylosing Spondylitis (WPAI-AS) Scale Scores and Bath Ankylosing Spondylitis Global Score (BAS-G) at Month 6 and 24
Description: WPAI-AS:6-question participant rated questionnaire to determine amount of absenteeism, presenteeism, work productivity loss, daily activity impairment due to AS for a period of 7 days prior to each visit. It yields 4 sub-scores: work time missed(absenteeism), impairment while working(presenteeism), overall work impairment(work productivity), activity impairment(daily activity impairment). These sub-scores are transformed to impairment percentages(range 0 to 100), with higher numbers indicating greater impairment, less productivity. BAS-G is used to indicate the effect of disease on participant's well-being. This scale is composed of 2 items ranging from 0 = very good to 10 =very bad. Total score ranges from 0 to 10: the higher the BAS-G score, the worse the participant's health status. Correlation coefficient between change from baseline in WPAI-AS and BAS-G score at Month 6, 24 was reported.
Time Frame: Month 6, Month 24
Population: as for outcome 6
Measure: Number; unit: Correlation coefficient
Arm/Group | Etanercept
Number analyzed (Participants) | 75
Correlation coefficient
  Month 6: Work Time Missed and BAS-G (n=55) | 0.34
  Month 6: Impairment While Working and BAS-G (n=44) | 0.56
  Month 6: Overall work impairment and BAS-G (n=38) | 0.55
  Month 6: Activity impairment and BAS-G (n=72) | 0.64
  Month 24: Work Time Missed and BAS-G (n=36) | 0.25
  Month 24: Impairment While Working and BAS-G(n=27) | 0.28
  Month 24: Overall work impairment and BAS-G (n=23) | 0.26
  Month 24: Activity impairment and BAS-G (n=56) | 0.60

15. Secondary Outcome: Correlation Between Work Productivity and Activity Impairment Questionnaire - Ankylosing Spondylitis (WPAI-AS) Scale Scores and 36-Item Short-Form Health Survey (SF-36) Physical Component Summary (PCS) Score at Baseline
Description: WPAI-AS:6-item questionnaire to determine amount of absenteeism,presenteeism,work productivity loss,daily activity impairment attributable to AS during 7 days prior to each visit.It yields 4 sub-scores:work time missed(absenteeism),impairment while working(presenteeism),overall work impairment(work productivity), activity impairment(daily activity impairment).Sub-scores transformed to impairment percentages(range 0 to 100), higher numbers=greater impairment,less productivity.SF-36:standardized survey evaluating 8 aspects of functional health,well being(physical,social functioning; physical,emotional role limitations; bodily pain; general health; vitality; mental health).8 aspects summarized as PCS and mental component summary (MCS).Scores normalized to United States population to have mean=50,standard deviation=10 (norm based scoring with <50=lower level of functioning and >50=higher level of functioning). Correlation coefficient between WPAI-AS and PCS score at baseline was reported.
Time Frame: Baseline
Population: as for outcome 7
Measure: Number; unit: Correlation coefficient
Arm/Group | Etanercept
Number analyzed (Participants) | 80
Correlation coefficient
  Work Time Missed and PCS (n=66) | -0.52
  Impairment While Working and PCS (n=54) | -0.52
  Overall work impairment and PCS (n=48) | -0.57
  Activity impairment and PCS (n=77) | -0.43

16. Secondary Outcome: Correlation Between Work Productivity and Activity Impairment Questionnaire - Ankylosing Spondylitis (WPAI-AS) Scale Scores and 36-Item Short-Form Health Survey (SF-36) Physical Component Summary (PCS) Score at Month 6 and 24
Description: WPAI-AS:6-item questionnaire to determine amount of absenteeism,presenteeism,work productivity loss,daily activity impairment attributable to AS during 7 days prior to each visit.It yields 4 sub-scores:work time missed(absenteeism),impairment while working(presenteeism),overall work impairment(work productivity),activity impairment(daily activity impairment).Sub-scores transformed to impairment percentages(range 0 to 100),higher numbers=greater impairment,less productivity.SF-36:standardized survey evaluating 8 aspects of functional health,well being(physical,social functioning; physical,emotional role limitations; bodily pain; general health; vitality; mental health).8 aspects summarized as PCS and MCS. Scores normalized to United States population to have mean=50,standard deviation=10 (norm based scoring with <50=lower level of functioning and >50=higher level of functioning). Correlation coefficient between change from baseline in WPAI-AS and PCS score at Month 6, 24 was reported.
Time Frame: Month 6, Month 24
Population: as for outcome 6
Measure: Number; unit: Correlation coefficient
Arm/Group | Etanercept
Number analyzed (Participants) | 75
Correlation coefficient
  Month 6: Work Time Missed and PCS (n=51) | -0.41
  Month 6:Impairment While Working and PCS (n=41) | -0.36
  Month 6: Overall work impairment and PCS(n=35) | -0.36
  Month 6: Activity impairment and PCS(n=66) | -0.57
  Month 24: Work Time Missed and PCS(n=28) | -0.52
  Month 24: Impairment While Working and PCS(n= 22) | -0.25
  Month 24: Overall work impairment and PCS(n= 18) | -0.36
  Month 24: Activity impairment and PCS (n=45) | -0.60

17. Secondary Outcome: Correlation Between Work Productivity and Activity Impairment Questionnaire - Ankylosing Spondylitis (WPAI-AS) Scale Scores and 36-Item Short-Form Health Survey (SF-36) Mental Component Summary Score (MCS) at Baseline
Description: WPAI-AS: 6-item questionnaire to determine amount of absenteeism, presenteeism, work productivity loss, daily activity impairment attributable to AS during 7 days prior to each visit. It yields 4 sub-scores: work time missed (absenteeism), impairment while working (presenteeism), overall work impairment (work productivity), activity impairment (daily activity impairment). Sub-scores transformed to impairment percentages (range 0 to 100), higher numbers=greater impairment,less productivity. SF-36:standardized survey evaluating 8 aspects of functional health, well being (physical, social functioning; physical, emotional role limitations; bodily pain; general health; vitality; mental health). 8 aspects summarized as PCS and MCS. Scores normalized to United States population to have mean=50, standard deviation=10 (norm based scoring with <50=lower level of functioning and >50=higher level of functioning). Correlation coefficient between WPAI-AS and MCS score at baseline was reported.
Time Frame: Baseline
Population: as for outcome 7
Measure: Number; unit: Correlation coefficient
Arm/Group | Etanercept
Number analyzed (Participants) | 80
Correlation coefficient
  Work Time Missed and MCS (n=66) | -0.06
  Impairment While Working and MCS (n=54) | -0.38
  Overall work impairment and MCS (n=48) | -0.41
  Activity impairment and MCS (n=77) | -0.51

18. Secondary Outcome: Correlation Between Work Productivity and Activity Impairment Questionnaire - Ankylosing Spondylitis (WPAI-AS) Scale Scores and 36-Item Short-Form Health Survey (SF-36) Mental Component Summary Score (MCS) at Month 6 and 24
Description: WPAI-AS:6-item questionnaire to determine amount of absenteeism,presenteeism,work productivity loss,daily activity impairment attributable to AS during 7 days prior to each visit.It yields 4 sub-scores:work time missed(absenteeism),impairment while working(presenteeism),overall work impairment(work productivity), activity impairment(daily activity impairment).Sub-scores transformed to impairment percentages(range 0 to 100), higher numbers=greater impairment,less productivity.SF-36:standardized survey evaluating 8 aspects of functional health,well being(physical,social functioning; physical,emotional role limitations; bodily pain; general health; vitality; mental health).8 aspects summarized as PCS and MCS. Scores normalized to United States population to have mean=50,standard deviation=10(norm based scoring with <50=lower level of functioning and >50=higher level of functioning). Correlation coefficient between change from baseline in WPAI-AS and MCS score at Month 6, 24 was reported.
Time Frame: Month 6, Month 24
Population: as for outcome 6
Measure: Number; unit: Correlation coefficient
Arm/Group | Etanercept
Number analyzed (Participants) | 75
Correlation coefficient
  Month 6: Work Time Missed and MCS (n=51) | -0.19
  Month 6: Impairment While Working and MCS(n=41) | -0.33
  Month 6: Overall work impairment and MCS(n=35) | -0.45
  Month 6: Activity impairment and MCS(n=66) | -0.29
  Month 24: Work Time Missed and MCS(n=28) | 0.038
  Month 24: Impairment While Working and MCS(n= 22) | -0.006
  Month 24: Overall work impairment and MCS(n= 18) | 0.36
  Month 24: Activity impairment and MCS(n=45) | -0.39

19. Secondary Outcome: Correlation Between Work Productivity and Activity Impairment Questionnaire - Ankylosing Spondylitis (WPAI-AS) Scale Scores and Euro Quality of Life-5 Dimensions (EQ-5D) Total Score at Baseline
Description: WPAI-AS:6-question participant rated questionnaire to determine amount of absenteeism, presenteeism, work productivity loss, daily activity impairment due to AS during 7 days prior to each visit. It yields 4 sub-scores: work time missed(absenteeism), impairment while working(presenteeism), overall work impairment(work productivity), activity impairment(daily activity impairment). These sub-scores are transformed to impairment percentages(range 0 to 100), with higher numbers=greater impairment, less productivity. EQ-5D:participant rated questionnaire to assess health-related quality of life in terms of single utility score. Health state profile component assesses level of current health for 5 domains: mobility,self-care,usual activities,pain/discomfort and anxiety/depression; Scale range 1 to 3 (1=better health state [no problems], 3=worst health state [confined to bed]). Correlation coefficient between WPAI-AS and EQ-5D total score at baseline was reported.
Time Frame: Baseline
Population: as for outcome 7
Measure: Number; unit: Correlation coefficient
Arm/Group | Etanercept
Number analyzed (Participants) | 80
Correlation coefficient
  Work Time Missed and EQ-5D (n=66) | -0.17
  Impairment While Working and EQ-5D (n=54) | -0.58
  Overall work impairment and EQ-5D (n=48) | -0.59
  Activity impairment and EQ-5D (n=78) | -0.52

20. Secondary Outcome: Correlation Between Work Productivity and Activity Impairment Questionnaire - Ankylosing Spondylitis (WPAI-AS) Scale Scores and Euro Quality of Life-5 Dimensions (EQ-5D) Total Score at Month 6 and 24
Description: WPAI-AS:6-question participant rated questionnaire to determine amount of absenteeism, presenteeism, work productivity loss, daily activity impairment due to AS during 7 days prior to each visit. It yields 4 sub-scores: work time missed(absenteeism), impairment while working(presenteeism), overall work impairment(work productivity), activity impairment(daily activity impairment). These sub-scores are transformed to impairment percentages(range 0 to 100), with higher numbers=greater impairment, less productivity. EQ-5D:participant rated questionnaire to assess health-related quality of life in terms of single utility score. Health state profile component assesses level of current health for 5 domains: mobility,self-care,usual activities,pain/discomfort and anxiety/depression; Scale range 1 to 3 (1=better health state [no problems], 3=worst health state [confined to bed]). Correlation coefficient between change from baseline in WPAI-AS and EQ-5D total score at Month 6, 24 was reported.
Time Frame: Month 6, Month 24
Population: as for outcome 6
Measure: Number; unit: Correlation coefficient
Arm/Group | Etanercept
Number analyzed (Participants) | 75
Correlation coefficient
  Month 6: Work Time Missed and EQ-5D (n=55) | -0.19
  Month 6: Impairment While Working and EQ-5D(n=44) | -0.60
  Month 6: Overall work impairment and EQ-5D(n=38) | -0.59
  Month 6: Activity impairment and EQ-5D(n=72) | -0.33
  Month 24: Work Time Missed and EQ-5D(n=34) | 0.007
  Month 24: Impairment While Working and EQ-5D(n=26) | -0.33
  Month 24: Overall work impairment and EQ-5D(n= 22) | -0.20
  Month 24: Activity impairment and EQ-5D(n=54) | -0.43

21. Secondary Outcome: Correlation Between Work Productivity and Activity Impairment Questionnaire - Ankylosing Spondylitis (WPAI-AS) Scale Scores and Euro Quality of Life (EQ-5D) Visual Analog Scale (VAS) Score at Baseline
Description: WPAI-AS:6-question participant rated questionnaire to determine amount of absenteeism, presenteeism, work productivity loss, daily activity impairment due to AS for a period of 7 days prior to each visit. It yields 4 sub-scores: work time missed(absenteeism), impairment while working(presenteeism), overall work impairment(work productivity), activity impairment(daily activity impairment). These sub-scores are transformed to impairment percentages(range 0 to 100), with higher numbers indicating greater impairment, less productivity. EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicate a better health state. Correlation coefficient between WPAI-AS and EQ-5D VAS score at baseline was reported.
Time Frame: Baseline
Population: as for outcome 7
Measure: Number; unit: Correlation coefficient
Arm/Group | Etanercept
Number analyzed (Participants) | 80
Correlation coefficient
  Work Time Missed and EQ-5D VAS (n=64) | -0.06
  Impairment While Working and EQ-5D VAS (n=54) | -0.42
  Overall work impairment and EQ-5D VAS (n=47) | -0.47
  Activity impairment and EQ-5D VAS (n=75) | -0.59

22. Secondary Outcome: Correlation Between Work Productivity and Activity Impairment Questionnaire - Ankylosing Spondylitis (WPAI-AS) Scale Scores and Euro Quality of Life (EQ-5D) Visual Analog Scale (VAS) Score at Month 6 and 24
Description: WPAI-AS:6-question participant rated questionnaire to determine amount of absenteeism, presenteeism, work productivity loss, daily activity impairment due to AS for a period of 7 days prior to each visit. It yields 4 sub-scores: work time missed(absenteeism), impairment while working(presenteeism), overall work impairment(work productivity), activity impairment(daily activity impairment). These sub-scores are transformed to impairment percentages(range 0 to 100), with higher numbers indicating greater impairment, less productivity. EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicate a better health state. Correlation coefficient between change from baseline in WPAI-AS and EQ-5D VAS score at Month 6, 24 was reported.
Time Frame: Month 6, Month 24
Population: as for outcome 6
Measure: Number; unit: Correlation coefficient
Arm/Group | Etanercept
Number analyzed (Participants) | 75
Correlation coefficient
  Month 6: Work Time Missed, EQ-5D VAS (n=53) | -0.15
  Month 6: Impairment While Working, EQ-5D VAS(n=44) | -0.57
  Month 6: Overall work impairment, EQ-5D VAS(n=38) | -0.62
  Month 6: Activity impairment, EQ-5D VAS (n=70) | -0.54
  Month 24: Work Time Missed, EQ-5D VAS (n=34) | 0.009
  Month 24:Impairment While Working, EQ-5D VAS(n=26) | -0.32
  Month 24: Overall work impairment, EQ-5D VAS(n=23) | -0.36
  Month 24: Activity impairment, EQ-5D VAS (n=53) | -0.52

ADVERSE EVENTS:
Description: Only serious adverse events (SAEs) were planned to be collected. Other AEs were not collected as per planned analysis for this non-interventional study.
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 0/80
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restriction Description: Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.